CLINICAL TRIAL: NCT07032636
Title: Reducing Crises and Suicide Within the Idaho Army National Guard - Enhancement of the First Line Leader Program
Brief Title: Reducing Crises and Suicide Within the Idaho Army National Guard
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Idaho Army National Guard (Unknown)
Responsible Party: Principal Investigator, Todd Bishop, Assistant Professor- Department of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00009623
Record Dates: First submitted 2025-05-27; First posted 2025-06-24 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Crisis Response Plan; Crisis Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FLL + TAP (Active Comparator): This will be a 1-day initial training that incorporates 12 leadership meetings, delivered during monthly drill weekends, and the FLLs will discuss program feasibility and acceptability with the program leadership. In addition to the standard FLL training, this group will learn about the Total Health Action Plan (TAP) and how to deploy it with their soldiers. The Investigators will measure fidelity of TAP delivery, soldier engagement and satisfaction rates, and whether NCOs are more responsive to soldiers reporting problems.
  Interventions: Behavioral: Crisis Intervention - The First Line Leaders (FLL) program will utilize templated guides developed with stakeholders from the Idaho Army National Guard (ARNG), known as the Total Health Action Plan (T
- FLL (Active Comparator): This is the existing 1-day initial training that incorporates 12 leadership meetings, delivered during monthly drill weekends currently being delivered by the Idaho Army National Guard. FLLs will discuss program feasibility and acceptability with the program leadership.
  Interventions: Behavioral: Crisis Intervention - The First Line Leaders (FLL) program will utilize templated guides developed with stakeholders from the Idaho Army National Guard (ARNG), known as the Total Health Action Plan (T
- No FLL (No Intervention): Participants assigned to this condition will receive training as usual and have not been assigned FLL training by the Idaho Army National Guard.

INTERVENTIONS:
Behavioral: Crisis Intervention - The First Line Leaders (FLL) program will utilize templated guides developed with stakeholders from the Idaho Army National Guard (ARNG), known as the Total Health Action Plan (T — The Investigators are developing training programs for soldiers and leaders to enhance their communication skills, problem-solving abilities, and approachability. They will be randomized to one of three different groups.
  Arms: FLL; FLL + TAP

SUMMARY:
Military suicide is an ongoing public health concern, particularly within the Army National Guard (ARNG), with longstanding effects on fellow soldiers, family, and friends. The straddling of military and civilian worlds for ARNG can worsen risk factors for suicide, including increased social isolation, disruption to family life, and employment difficulties. One promising framework that addresses both unit cohesion and social support is the First Line Leaders (FLL) program, recently designated by ARNG for nation-wide dissemination. The program is centered on enhancing the relationship between junior enlisted soldiers (JES) and their assigned non-commissioned officer (NCO). The Investigators propose to study an augmented FLL program that includes templated guides developed in collaboration with Idaho ARNG stakeholders. The guides, referred to as TAP (Total Health Action Plan), were adapted from two empirically based interventions, Crisis Response Planning and Problem-Solving Therapy, and consist of prompts for open communication and effective engagement and guidelines for responding to impending or current behavioral distress. Given their elevated suicide risk, the Idaho ARNG is a crucial setting to develop this upstream intervention.

In this study, the Investigators propose to compare the augmented FLL + TAP program to FLL only, and training as usual (n= 50 NCOs and 100 JES per group) with quarterly assessments for up to one year. The Investigators will examine a random selection of deidentified counseling templates to examine the type and frequency of counseling sessions involving acute crisis and behavioral health difficulties, and online ratings from a random selection of JES using validated instruments to assess upstream indicators of behavioral distress and suicide risk and resilience. The Investigators will also conduct qualitative interviews with a random selection of 20% of the NCOs (n = 30) and JES (n = 60) enrolled in the project to provide personalized perspectives of program experiences.

The Investigators propose three aims to guide this research. (1) Collaborate with Idaho ARNG stakeholders to integrate TAP into FLL programming via: a) development and refinement of TAP training materials, b) building templated counseling statements that align with FLL and TAP, and c) education of Idaho ARNG training cadre in the delivery of TAP. (2) Evaluate fidelity, feasibility, and acceptability of FLL and FLL + TAP through a mixed methods approach of qualitative interviews with FLLs and JESs and evaluation of data from templated counseling sessions. (3) Examine the impact of FLL+TAP versus FLL versus training as usual on unit morale, cohesion, and general functioning.

ELIGIBILITY:
Inclusion Criteria:

* Enlistment or commission in the Idaho ARNG at the time of enrollment
* Age 18 or greater
* Ability to complete all study questionnaires and interview procedures
* Has at least one year remaining on National Guard contract

Exclusion Criteria:

- Less than one year remaining on their contract with the National Guard

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in Fidelity to TAP. | Baseline, Month 3, Month 6, Month 9, and, Month 12.
  Fidelity to TAP will be assessed by examining counseling statements where an intervention was completed on the templated counseling statement forms generated by our Stakeholder Advisory Board (SAB) using a Likert-type scale (e.g., 1 = poor fidelity, 5 = excellent fidelity). The total range of possible scores is from 1 to 5, with higher scores indicating better fidelity.
Estimate of TAP usage at Follow-Up Assessments | Baseline, Month 3, Month 6, Month 9, and Month 12
  Participants will be asked to complete a survey item assessing how many times they used a TAP during the 3-, 6-, 9-, and 12-month follow-up visits. Response options will range from 0 to 99. The higher the score, the more TAPs the participant estimates they used during the given assessment period.
Mean satisfaction with TAP while in the FLL training program | Baseline, Month 3, Month 6, Month 9, and, Month 12
  Participants will be asked to complete a survey called Client Satisfaction Questionnaire (CSQ). CSQ items are rated on a Likert-type scale that ranges from 0 to 4, with the higher total score indicating greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bishop, PhD, Principal Investigator — University of Rochester
Locations (1):
- Idaho Army National Guard, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No